CLINICAL TRIAL: NCT03717363
Title: Efficacy of Training Programme in Physical Activity Promotion in Patients With High Risk of Cardiovascular Disease
Brief Title: Training Programme in Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Principal Investigator, Felicitas Garcia, Principal Investigator. Head of cardio-respiratory rehabilitation unit., Hospital Mutua de Terrassa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A2_2014
Record Dates: First submitted 2018-10-05; First posted 2018-10-24 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Cardiovascular Risk Factor; Cardiovascular Disease
Keywords: Training Programme; Physical Activity; cardiovascular primary prevention
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: randomitzed interventional study with control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Educational talk: an educational talk given by the nurse and the physiotherapist about the components of a cardiosaluble lifestyle.
  Interventions: Behavioral: Educational talk
- Interventional group (Experimental): Training program in the primary care center supervised by a physiotherapist. The duration is two months and the frequency of sessions 3 times / week. Each session lasts 60 minutes.(30 minutes of aerobic exercise and 15 minutes of strength exercise).
  Interventions: Procedure: Training programme; Behavioral: Educational talk

INTERVENTIONS:
Procedure: Training programme — Training program in the primary care center supervised by a physiotherapist. The duration is two months and the frequency of sessions 3 times / week. Each session lasts 60 minutes.(30 minutes of aerobic exercise and 15 minutes of strength exercise).
  Arms: Interventional group
Behavioral: Educational talk — An educational talk given by the nurse and the physiotherapist about the components of a cardiosaluble lifestyle.

SUMMARY:
The primary prevention of cardiovascular disease is an unresolved health problem. A sedentary lifestyle and a low cardiorespiratory condition both increase the risk of cardiovascular disease, at a similar extent as that promoted by traditional risk factors, such as smoking, high blood pressure or dyslipidemia. The scientific evidence regarding the effect of the promotion of an active lifestyle on primary cardiovascular prevention is limited. Several studies have shown that structured training programs (TP) are effective at short term, but at the medium or long term their efficacy is still unknown. There are very few randomized controlled trials, and there are almost no studies conducted in the primary care setting which analyze the long-term effects of this type of program on primary cardiovascular prevention. The investigators performed in primary care a previous quasi-experimental study without control group demonstrating the short-term effectiveness in the improvements of both physical condition and in the practice of physical exercise of this TP, the shortest so far analyzed in primary care. With the current study the investigators also want to demonstrate its short-term efficacy in the promotion of moderate-high physical activity and in the practice of physical exercise, through a high-evidence design such as a randomized clinical trial with a control group, also the extension of such efficacy in the medium and long term.

Objective:

To determine the efficacy of a supervised 2 month TP on short-term (1 month post-TP), medium-term (6 months post-TP) and long-term (12 months post-TP) promotion of moderate-high physical activity and practice of physical exercise, in a sedentary population with high cardiovascular risk, attending primary care centres.

Methodology:

A parallel, randomized, intervention study, with a control group. Inclusion criteria: Men and women of an age between 35 and 70 years, attending a primary care center in hospital reference area, with high cardiovascular risk. Sedentary lifestyle defined by a score <2 in the brief Physical Activity Questionnaire for care consultations primary adapted to measure the frequency of physical exercise and with a total result in the International Physical Activity Questionnaire (IPAQ)-long version ≤1500 METs x minutes/week, who agree to participate and commit to compliance with the program.

Participants were randomized (automated list generation) to a control group, consisting in conventional management or to an intervention group (TP 2 months, 3 times / week). Both groups received an educational talk about cardiovascular risk, healthy diet habits and cardio-healthy exercise at the beginning of TP. Assessments were performed at baseline, and at 3, 8 and 14 months.

OUTCOMES:

1. Main outcome measure: differences between groups in the proportion of participants with an "Effective response in Physical Activity ". This effective response was considered if there was an increase ≥ 240 METs x minutes / week in the moderate-high physical activity (measured by IPAQ-long version) in the final evaluation.
2. Secondary outcome variables: differences between groups in the change in:

   1. Physical exercise: quantitatively (measured by the sum of the results obtained in items 22-25 of the IPAQ-long version), frequency (Physical Activity Questionnaire for care consultations primary adapted to measure the frequency of physical exercise), and intention (Questionnaire of Stages of Change of Exercise (QSCE)-Short Form).
   2. Global physical activity (measured with the total result in the IPAQ-long version).
   3. Physical condition: ergometric variables (Peak Oxygen Consumption, exercise duration, anaerobic threshold moment)) and 6 Minute Walk Test.
3. Other efficacy and safety variables: differences between groups in the changes in:

   1. Anthropometric variables.
   2. Blood pressure.
   3. Biochemical parameters.
   4. Mediterranean diet (simplified version of the questionnaire ¨Adherence to the Mediterranean Diet¨).
   5. Quality of life (questionnaire SF36-long version).
   6. Mood (Beck depression index).

DETAILED DESCRIPTION:
INTRODUCTION The primary prevention of cardiovascular disease (CVD), the main cause of morbidity and mortality in most Western countries, is a priority. A sedentary lifestyle and a low cardiorespiratory condition increase the risk of CVD with the same impact as the presence of Cardiovascular Risk Factors (CVRF) such as smoking, high blood pressure or dyslipidemia.

Among the interventions aimed at promoting Physical Activity (PA), there are supervised Training Programs (TP). In Primary Cardiovascular Prevention (PCVP), supervised TP appear to be effective in the short term in improving cardiorespiratory fitness, glycemic control, cardiovascular (CV) risk profile and in promoting a more active lifestyle. The effect of these TPs in the medium-long term in PCVP is still unknown. In primary care, the ideal context in which to apply interventions aimed at the promotion of a cardio-healthy lifestyle, the few randomized controlled trials (RCT) conducted on the effects of this type of interventions in the medium-long term obtain contradictory results.

The investigators aims to analyze the short, medium and long term efficacy of a supervised TP, performed in primary care and with the shortest duration so far contemplated (2 months), in the promotion of moderate-high PA and in practice of physical exercise, in a sedentary population with high CV risk.

OBJECTIVES:

1. Main objective: To determine the short, medium and long term efficacy in the field of primary care of a supervised TP in the promotion of moderate-high PA, measured with the variable " Effective response in PA " that is defined as an increase in moderate-high PA (measured by the sum of the results in the moderate PA dimension and vigorous PA dimension of the International Physical Activity Questionnaire (IPAQ)-long version of at least 240 METs x minute/week (METs x min/wk), in a sedentary population with high CV risk .
2. Secondary objectives: Determine the short, medium and long term efficacy in the primary care area of a supervised TP in:

   1. The practice of regular physical exercise, measured with items 22-25 of the IPAQ-long version, with the Short Physical Activity Questionnaire for Primary Care Consultations (PAQCCP) adapted to measure the frequency of exercise and with the Questionnaire of Stages of Change of Exercise-Short Form (QSCE-Short form).
   2. The overall PA measured with the total result obtained in the IPAQ-long version.
   3. The cardiorespiratory condition measured with the Six Minute Walking Test (6MWT) and the Cardiopulmonary Exercise Testing (CPET) variables Peak Oxygen Consumption (VO2peak), exercise duration and Anaerobic Threshold (AT) moment.
   4. The evolution of the main CVRF (smoking, body mass index, abdominal circumference, systolic and diastolic blood pressure, glycaemia, glycated haemoglobin, total cholesterol, high-density lipoprotein cholesterol (hdl-c), low-density lipoprotein cholesterol (ldl-c), triglycerides) and in the composition of the diet measure with the simplified version of the questionnaire ¨Adherence to the Mediterranean Diet¨.
   5. The quality of life quantified with the questionnaire SF36-long version and in the state of mind with the Beck Depression Index.

METHODOLOGY

DESIGN: Randomized controlled trial.

SUBJECTS, SCOPE AND CRITERIA FOR INCLUSION TO THE STUDY: Participants aged 35 to 70 years old from the ¨Rambla¨ primary care center in the reference area of the Mutua Terrassa University Hospital, sedentary and with high CV risk who agreed to participate and were committed to a fulfillment of the program.

Sedentary was considered one with a score in the PAQCCP (Puig A et al., Aten Primaria 2012; 44 (8): 485-93), adapted to measure the frequency of physical exercise, less than 2 and with a result in the total IPAQ-long version ≤1500 METs x min /wk.

The high CV risk was defined by the presence of any of the following conditions: Diabetes Mellitus type 2; Metabolic syndrome, defined by the criteria of the National Cholesterol Education Program (NCEP) / American Heart Association (AHA); and / or Hypertension with at least one associated CVRF (smoking, dyslipidemia, obesity).

EXCLUSION CRITERIA: Last ambulatory visit performed in a period greater than one year at the time of inclusion, pregnant women, comorbidities that prevent the patient from doing the TP, not autonomy for a commitment to program compliance and / or previous CV events.

STUDY PERIOD: after the inclusion period and the completion of an educational talk, the participants were followed a total of 14 months. The total duration of the study was 36 months to complete all the groups and their follow-up.

SAMPLING AND TOTAL SIZE:

Accepting an alpha risk of 0.05 and a beta risk of 0.20 in a bilateral contrast, 73 participants in the control group and 73 in the intervention group were required to detect a clinically relevant difference between groups of at least 20% in the proportion of participants with "Effective response in PA". This response has been defined as the increase in the moderate-high PA measured with the sum of the results in the moderate PA dimension and vigorous PA dimension of the IPAQ-long version, of minimum 240 METs x min /wk. A proportion of responding participants was assumed in PA of 11% in the control group and 31% in the intervention group. A follow-up loss rate of 15% was estimated. The ARCOSENO approach was used.

Sampling was carried out by a simple randomization in an automated way, assigning to the participants an identifier number corresponding to the control or intervention group.

PROCEDURE, INSTRUMENTATION AND COLLECTION OF INFORMATION:

The family doctor of the primary care center made a first selection of candidates. After receiving all the necessary information about the study and signing the informed consent, the family doctor referred participants to the rehabilitation doctor. In the initial assessment of the rehabilitation doctor a socio-demographic, anthropometric, analytical variables (haemoglobin, lipid profile, glycemia, glycated haemoglobin and creatinine), systolic and basal diastolic blood pressure, baseline heart rate, pathological history and CVRF and pharmacological treatment were collected. In addition, the PAQCCP, the QSCE-Short Form, the IPAQ-long version and the Beck Depression Index. All the questionnaires used in the study were translated and validated into Spanish. 6MWT and CPET were performed. If the CPET was clinically and /or electrically positive, the participants was not included in the study until it was assessed by the Cardiologist of the program, and the latter would rule out the presence of established CVD. After the assessment, the inclusion in the study of the selected participants was confirmed and they were assigned to the control group or intervention group as it corresponded to the automated randomization.

If the participant was assigned to the intervention group he received the following attention:

* An educational talk about CV risk, diet and cardio-healthy exercise, given by the nurse and the physiotherapist. The nurse gave the participant the information leaflet on heart-healthy lifestyles and administered the simplified version of the questionnaire ¨Adherence to the Mediterranean Diet¨ and the SF36 questionnaire-long version.
* Control visit by nurse, family doctor and rehabilitation doctor per month, at 6 months and 12 months post-TP (coinciding in time with 3, 8 and 14 months of the day of the educational talks common to the control group). In each visit the same variables were collected as in the initial assessment and also possible pharmacological changes, incidences, consultations with Cardiologist and medical tests performed.

If the participant was assigned to the control group, he received the same attention as the intervention group except that he did not perform the TP. The controls by nursing, family doctor and rehabilitation doctor were carried out at 3, 8 and 14 months of the day of the educational talks.

An action protocol was followed for the control group and for the intervention group, so that in the event that during the follow-up the CPET was clinically and / or electrically positive, it was evaluated by the Cardiologist and if established CVD was confirmed, the participant left the study.

VARIABLES:

1. Variable main result: differences between groups in the percentage of participants that achieve an " Effective response in PA " defined by an increase in moderate-high PA measured with the sum of the results in the PA dimension moderate and vigorous PA dimension of the IPAQ-long version, of minimum 240 METs x min / wk.
2. Secondary outcome variables: differences between groups in the changes in the amount of physical exercise measured by the sum of the results obtained in items 22-25 of the IPAQ-long version, in the frequency of physical exercise (PAQCCP adapted), and in the exercise intention (QSCE-Short form), changes in the global PA measured with the total result in the IPAQ-long version, change in the physical condition variables (ergometric variables (VO2peak, exercise duration, AT moment) and 6MWT).
3. Other secondary variables: differences between groups in the changes in the analytical and anthropometric variables, in blood pressure, in the simplified version of the questionnaire ¨Adherence to the Mediterranean Diet¨, in the questionnaire SF36-long version and in the Beck Depression Index.

DATA ANALYSIS:

After collecting the variables, the data has been entered into a relational Access database designed ad-hoc.

At this moment the debugging, consistency and quality control of the data are being carried out, together with the first statistical analyzes at the post-program month (3 months post-talks) through the Stata vs 13.0 program.

The comparison of results between control group and intervention group will be made at 3, 8 and 14 months of the day of the talks.

ELIGIBILITY:
Inclusion Criteria:

* From a primary care center in the reference area of our hospital
* High cardiovascular risk
* Sedentary defined by a score in the brief Physical Activity Questionnaire for primary care consultations (CAFBCAP) adapted for measure the frequency of physical exercise <2 and with a result in the IPAQ-total long version ≤1500 METsxmin / week
* they accept to participate and commit to compliance with the program.

Exclusion Criteria:

* Last ambulatory visit more than a year ago
* Pregnant women
* Comorbidities that make the patient unable to do the programme or to be dependen on second person for journeys
* Previous cardiovascular events.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Difference between groups in the proportion of patients who achieve the ¨Effective response in Physical Activity¨ | 1 month post intervention; 6 months post intervention and 12 months post intervention
  The ¨Effective response in Physical Activity¨ is defined as an minimum increase of 240 METsxmin / wk in moderate-vigorous Physical Activity measured with the sum of the results in the moderate and vigorous Physical Activity dimension of the International Physical Activity Questionnaire-Long version.
  The International Physical Activity Questionnaire- long version (27 items) collects data in different domains and intensities (moderate, vigorous,walking) and includes sitting time. The units of measurement are METsxmin/week. The amount of physical activity is recorded by intensity (moderate, vigorous, walking) and the amount of total physical activity obtained by adding the records in each dimension according to intensity . A category of low physical activity is considered a result in the total physical activity below 600 METsxmin / week, moderate between 600 and 3000 METsxmin / week and high above 3000 MEtsxmin / week.

CONTACTS AND LOCATIONS:
Overall Officials: Felicitas García Ortún, MD, Principal Investigator — Fundación Asistencial MutuaTerrassa
Locations (1):
- Hospital Universitari Mutua Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boule NG, Kenny GP, Haddad E, Wells GA, Sigal RJ. Meta-analysis of the effect of structured exercise training on cardiorespiratory fitness in Type 2 diabetes mellitus. Diabetologia. 2003 Aug;46(8):1071-81. doi: 10.1007/s00125-003-1160-2. Epub 2003 Jul 10. PMID 12856082
- [Result] Eriksson KM, Westborg CJ, Eliasson MC. A randomized trial of lifestyle intervention in primary healthcare for the modification of cardiovascular risk factors. Scand J Public Health. 2006;34(5):453-61. doi: 10.1080/14034940500489826. PMID 16990155
- [Result] Balducci S, Zanuso S, Nicolucci A, De Feo P, Cavallo S, Cardelli P, Fallucca S, Alessi E, Fallucca F, Pugliese G; Italian Diabetes Exercise Study (IDES) Investigators. Effect of an intensive exercise intervention strategy on modifiable cardiovascular risk factors in subjects with type 2 diabetes mellitus: a randomized controlled trial: the Italian Diabetes and Exercise Study (IDES). Arch Intern Med. 2010 Nov 8;170(20):1794-803. doi: 10.1001/archinternmed.2010.380. PMID 21059972
- [Derived] Garcia-Ortun F, Jaen A, Sola L, Gonzalez-Gil L, Garreta R, de la Sierra A. Physical training program for people at risk of cardiovascular disorders in the primary care setting: A randomized clinical trial. Med Clin (Barc). 2022 Nov 25;159(10):475-482. doi: 10.1016/j.medcli.2022.01.020. Epub 2022 Mar 19. English, Spanish. PMID 35318946